CLINICAL TRIAL: NCT01970787
Title: A Trial of Radiofrequency Ablation for Anal Intraepithelial Neoplasia Using the HALO Ablation System
Acronym: AIN
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medtronic - MITG (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: B-250
Record Dates: First submitted 2013-10-22; First posted 2013-10-28 (Estimated); Results first posted 2016-07-14 (Estimated); Last update posted 2017-02-06 (Estimated); Status verified 2016-12

CONDITIONS: HIV-negative Subjects With Intra-anal Intraepithelial Neoplasia Containing High-Grade Squamous Intraepithelial Lesions
MeSH Terms: interventions — Radiofrequency Ablation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- RFA (Experimental): Assess the feasibility, safety, and efficacy of RF to the anal canal using the HALO Ablation System to eradicate anal HSIL lesions
  Interventions: Device: Radiofrequency Ablation (RFA) using the HALO Ablation System

INTERVENTIONS:
Device: Radiofrequency Ablation (RFA) using the HALO Ablation System
  Other Names: Barrx Ablation System

SUMMARY:
This is a Single-center prospective pilot trial involving up to 22 subjects. This study will assess the feasibility, safety, and efficacy of radiofrequency ablation (RFA) to the anal canal using the FDA cleared HALO Ablation System to eradicate anal HSIL lesions in HIV-negative subjects with intra-anal intraepithelial neoplasia (AIN). The study intervention will demonstrate that a reasonable proportion of subjects will be histologically cleared of their anal HSIL within the ETZ in a tolerable and relatively safe manner

ELIGIBILITY:
Inclusion Criteria:

* Age 18-75 years
* HRA 2 to 12 weeks prior to the 0 month RFA visit yielding one or more flat, non-condylomatous biopsy-proven HSILs that are

  1. Located entirely within in the eligible treatment zone
  2. Contiguous with the squamocolumnar junction Eligible treatment zone (ETZ) is defined as

  <!-- -->

  1. 3 cm above the dentate line to the anocutaneous line
  2. Half of the anorectal circumference (meaning no more than two contiguous quadrants)
* If female of child-bearing age, negative pregnancy test within 8 weeks of the 0 month RFA visit and declared intent to remain on birth control throughout the trial, or, declaration of infertility defined as subject report of status as post-menopausal or surgically sterile (status post hysterectomy or tubal ligation).
* HIV negative, ELISA/Western blot test obtained within 12 weeks of the 0 month RFA visit

Exclusion Criteria:

1. Any biopsy-proven HSIL entirely outside of the ETZ
2. Any biopsy-proven HSIL partially within the ETZ (for example, an HSIL lesion with extension to the perianal skin)
3. Any condylomas in the eligible treatment zone > 1/2 cm diameter

   • Note: Condylomas in the eligible treatment zone < 1/2 cm in diameter must be excised or cauterized (not treated topically or with IRC) before or during Visit 1 (0 month RFA visit)
4. Any anal or rectal pathology requiring treatment including ulcer, fistula, fissure, stenosis or proctitis
5. History of or present anal or rectal cancer
6. History of pelvic radiation therapy
7. History of HPV vaccination or plans to initiate HPV vaccination during the trial
8. History of ablation or resection therapy within the ETZ other than cauterization or excision of condyloma(s)
9. History of topical therapy (Imiquimod, 5-FU) within 6 months prior to the 0 month RFA visit within the ETZ
10. Hemorrhoids > grade II
11. Fecal incontinence (that the investigator feels may impair healing)
12. Concurrent disease requiring systemic immunosuppression therapy
13. Concurrent malignancy requiring systemic therapy
14. Life expectancy < 2 years

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2013-03; Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Laser Surgery Center, New York, New York, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- RFA Treatment: Assess the feasibility, safety, and efficacy of RF to the anal canal using the HALO Ablation System to eradicate anal HSIL lesions
  Radiofrequency Ablation (RFA) using the HALO Ablation System
Period: Overall Study
Arm/Group | RFA Treatment
Started | 22
Completed | 21
Not Completed | 1

BASELINE CHARACTERISTICS:
Population: HIV-negative subjects with AIN containing HSIL located within half of the anorectal circumference, which is defined as no more than two contiguous quadrants and in the study referred to as the eligible treatment zone (ETZ).
Arm/Group | RFA Treatment
Number analyzed (Participants) | 21
Age, Continuous [Mean (Full Range); unit: years] | 45 [32 to 65]
Gender [Count of Participants; unit: Participants]
  Female | 3
  Male | 18
Region of Enrollment [Number; unit: participants]
  United States | 21

OUTCOME MEASURES:

1. Primary Outcome: Clearance of Anal HSIL (High Grade Squamous Intraepithelial Lesion (HSIL)
Description: Participants with histologic clearance of anal HSIL within the ETZ (eligible treatment zone) at 12 months from first RFA treatment
Time Frame: 12 months
Measure: Number; unit: participants w histological clearance
Arm/Group | RFA Treatment
Number analyzed (Participants) | 21
participants w histological clearance | 19

2. Secondary Outcome: Feasibility and Ease of Technique
Description: Technical feasibility of applying RFA to the anal canal. Physician's assessment of ablation as optimal (complete ablation) versus sub-optimal (incomplete ablation)in the affected area in the anal canal.
  Data not collected and could not be analyzed
Time Frame: 12 months
Arm/Group | RFA Treatment
Number analyzed (Participants) | 0

3. Secondary Outcome: Tolerability
Description: Subject tolerability of the RFA procedure as measured by severity. Mild: Awareness of signs and symptoms, but easily tolerated; are of a minor irritant type; causing no loss of time from normal activities; symptoms would not require medication or a medical intervention; asymptomatic lab findings; marginal clinical relevance; signs and symptoms are transient.
  Moderate: Discomfort severe enough to cause interference with usual activities; minimal intervention.
  Severe: Incapacitating with inability to do work or usual activities; signs and symptoms may be of systemic nature or require medical evaluation or treatment.
Time Frame: 12 months
Measure: Number; unit: participants
Arm/Group | RFA Treatment
Number analyzed (Participants) | 21
participants
  bleeding associated with bowel movements | 20
  anal bleeding without a bowel movement, mild | 12
  anal bleeding without a bowel movement, moderate | 7
  severe bleeding associated with a bowel movement | 1

4. Secondary Outcome: Adverse Events
Description: Any related adverse event occuring in patients enrolled in this study. Event type and relationship to the device or procedure will be measured.
Time Frame: 12 months
Measure: Number; unit: participants
Arm/Group | RFA Treatment
Number analyzed (Participants) | 21
participants | 2

5. Secondary Outcome: Progression of HSIL to Cancer
Description: Histologic progression of HSIL to cancer as measured in biopsies read at the central pathology lab. Data not collected and could not be analyzed.
Time Frame: 12 months
Arm/Group | RFA Treatment
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Arm/Group | RFA Treatment
Serious Adverse Events (participants affected / at risk) | 0/21
Other Adverse Events (participants affected / at risk) | 2/21
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | RFA Treatment (N=21)
Anal pocket with purulent discharge (Injury, poisoning and procedural complications) | 1 (1)
Fever (Injury, poisoning and procedural complications) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less